CLINICAL TRIAL: NCT00665691
Title: Pilot Test for a Newly Developed Nutrition Screening Method: Pediatric Subjective Global Assessment
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PEDSGA
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2011-06

CONDITIONS: Compare Two Nutrition Screening Tools
Keywords: All Malignancies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Nutritional Screening Tools

INTERVENTIONS:
Other: Nutritional Screening Tools — To compare the nutrition risk identification abilities of two nutrition screening tools: PEDSGA tool and the standard assessment tool.

SUMMARY:
Researchers are studying ways to predict if cancer patients are at risk for poor nutrition during their chemotherapy treatment. They hope to identify children with nutrition problems early in treatment. This may help prevent weight loss and other nutrition problems later in treatment.

DETAILED DESCRIPTION:
The PEDSGA is a newly developed nutrition tool that includes a training manual that be used to teach health care professionals to identify at-risk patients by doing a nutrition physical exam. The PEDSGA also includes questions that the patient/caregiver answers regarding appetite, recent treatment, and activity level. This method of screening is new and may be able to identify at-risk patients better than the standard method. This study will use both methods and evaluate the two, in hope of determining which method works best to identify at-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* St. Jude Children's Research Hospital patient between 2 and 16 years of age who is actively receiving treatment for a hematologic or solid tumor malignancy
* Patient is not admitted to the transplant service
* Patient is able to read English or Spanish

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participant is between 2 and 16 years of age and receiving treatment for a hematologic or solid malignancy at St. Jude Children's Research Hospital.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2003-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To compare the ability of two nutrition screening tools to identify nutritionally at risk patients | Within 90 days of study completion

CONTACTS AND LOCATIONS:
Overall Officials: Karen Smith, RD, MS, LDN, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org/stjude/v/index.jsp?vgnextoid=f2bfab46cb118010VgnVCM1000000e2015acRCRD